CLINICAL TRIAL: NCT03212495
Title: Comparison Between Intra-articular Dexmedetomidine and Neostigmine as Adjuvant Analgesics After Knee Arthroscopy
Brief Title: Intra-articular Dexmedetomidine Versus Neostigmine After Knee Arthroscopy (a Comparative Study)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Mohammed AboelFadl, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: dexmedetomidine vs neostigmine
Record Dates: First submitted 2017-07-07; First posted 2017-07-11 (Actual); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Knee Injuries
Keywords: knee arthroscopy; dexmedetomidine; neostigmine
MeSH Terms: conditions — Knee Injuries | interventions — Dexmedetomidine; Neostigmine

STUDY DESIGN:
Intervention Model Description: Patients will be randomly allocated to one of two groups each including 50 patients; the group received either intraarticular dexametomidine or neostigmine .
Who Masked: Participant, Care Provider
Masking Description: , Patients were randomly allocated (using random table assignment) into two groups to receive one of the following intra-articular solutions (prepared by an individual not involved in the study) which were injected into the knee joint through the cannular sheath after withdrawal of camera, by the orthopaedic surgeon (who was also unaware of the nature of the study drugs) before the arthroscope removed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dexmedetomidine (D group) (Active Comparator): intraarticular administration of dexmedetomidine at the end of surgery
  Interventions: Drug: dexamedetomidine
- neostigmine (N group) (Active Comparator): intraarticular administration of neostigmine at the end of surgery.
  Interventions: Drug: neostigmine

INTERVENTIONS:
Drug: dexamedetomidine — intraarticular injection of 1µg/kg dexametomidine +18ml 0.25%bubivacaine in a total volume of 20 ml.
  Other Names: precedex; dexamedetomidine Hcl injection
  Arms: dexmedetomidine (D group)
Drug: neostigmine — intraarticular injection of 0.5mg/dose neostigmine +18ml 0.25%bubivacaine in a total volume of 20 ml.
  Other Names: prostigmine
  Arms: neostigmine (N group)

SUMMARY:
Knee arthroscopy is a minimally invasive day case procedure which may be done for diagnosis, meniscectomy or debridement. Arthroscopic surgery is associated with a variable degree of postoperative pain, which is caused by an irritation of free nerve endings of the synovial tissue, anterior fat pad, and joint capsule due to surgical excision and resection

DETAILED DESCRIPTION:
Many studies were done using different intra-articular agents as local anesthetics, opioids, ketamine and alfa2- adrenergic agonists for prevention and treatment of pain after knee surgeries.

Dexmedetomidine is a potent and highly selective alfa2-adrenoreceptor agonist. It has sedative-hypnotic, anxiolytic, analgesic, anesthetic and sympatholytic effects. Intra-articular dexmedetomidine was used in several studies to enhance postoperative analgesia after knee arthroscopy with an increased time to first analgesic request and a decreased need for postoperative analgesia Neostigmine is an anticholinesterase and also has antinociceptive effects when administered intrathecally or peripherally.

ELIGIBILITY:
Inclusion Criteria:

* patients aged above 18 years
* scheduled for elective arthroscopic knee surgery under intrathecal anaesthesia

Exclusion Criteria:

* Absolute or relative contraindications for intrathecal anaesthesia,
* Allergy for the studied drugs.
* Patients having history of cardiovascular, cerebrovascular, and respiratory diseases,
* Patients receiving chronic pain treatment or hypertension treated with alfa methyldopa, clonidine or beta adrenergic blockers were excluded from the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
postoperative pain | 36 hours after the end of the surgery.
  visual analogue pain scale

SECONDARY OUTCOMES:
nausea,vomiting | 36 hours after the end of the surgery.
  nausea and vomiting scales
sedation | 36 hours after the end of the surgery.
  Ramsay sedation score

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut governorate, Asyut, Egypt

REFERENCES:
- [Result] Al-Metwalli RR, Mowafi HA, Ismail SA, Siddiqui AK, Al-Ghamdi AM, Shafi MA, El-Saleh AR. Effect of intra-articular dexmedetomidine on postoperative analgesia after arthroscopic knee surgery. Br J Anaesth. 2008 Sep;101(3):395-9. doi: 10.1093/bja/aen184. Epub 2008 Jun 20. PMID 18567675
- [Result] Bondok RS, Abd El-Hady AM. Intra-articular magnesium is effective for postoperative analgesia in arthroscopic knee surgery. Br J Anaesth. 2006 Sep;97(3):389-92. doi: 10.1093/bja/ael176. Epub 2006 Jul 11. PMID 16835255
- [Result] Ebert T, Maze M. Dexmedetomidine: another arrow for the clinician's quiver. Anesthesiology. 2004 Sep;101(3):568-70. doi: 10.1097/00000542-200409000-00003. No abstract available. PMID 15329580